CLINICAL TRIAL: NCT01658436
Title: A Multicenter, Two Stage, Phase II Study, Evaluating the Efficacy of Oral BEZ235 Plus Best Supportive Care (BSC) Versus Placebo Plus BSC in the Treatment of Patients With Advanced Pancreatic Neuroendocrine Tumors (pNET) After Failure of mTOR Inhibitor Therapy.
Brief Title: BEZ235 Phase II Trial in Patients With Advanced Pancreatic Neuroendocrine Tumors (pNET) After Failure of mTOR Inhibitor Therapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBEZ235F2201; 2012-000675-16 (EudraCT Number)
Record Dates: First submitted 2012-07-06; First posted 2012-08-07 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Pancreatic Neuroendocrine Tumors (pNET)
Keywords: advanced pancreatic neuroendocrine tumor; BEZ235; pNET
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive | interventions — dactolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BEZ235 300 mg/400 mg bid (Stage 1) (Experimental): Stage 1 consisted of a single arm where patients received BEZ235 300mg or 400mg bid. Initially the study started with a dose of 400mg bid. However, following an amendment after the preliminary safety and tolerability data from the first 3 patients treated at the 400mg dose, the dosage was changed to 300mg bid.
  Interventions: Drug: BEZ235 (Stage 1)

INTERVENTIONS:
Drug: BEZ235 (Stage 1) — The investigational study drug used in this trial was BEZ235, which was supplied as 50mg, 200mg, 300mg, and 400mg solid dispersion sachets. Supply as 200mg and 50mg were provided for dose reduction. Patients were instructed to take the contents of one sachet of BEZ235 twice a day in the morning within 30 minutes after a light meal (breakfast).

SUMMARY:
This is a Phase II study in 2 stages, evaluating BEZ235 plus best supportive care (BSC) versus placebo plus BSC in patients with advanced pancreatic neuroendocrine tumors (pNET) after failure of mTOR inhibitor therapy.

Study design: This was a Phase II, two-stage, multicenter study, where Stage 1 was a single arm, open label design and Stage 2 was planned to be a randomized, double-blind study.

However, at the end of Stage 1, the futility was met and hence the Stage 2 was not initiated.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or metastatic, histologically confirmed low or intermediate grade pancreatic neuroendocrine tumor with radiological evidence of disease progression since last treatment
* Refractory disease to treatment with mTOR inhibitor
* Measurable disease per RECIST Version 1.1 using Computed Tomography (CT) or Magnetic Resonance Imaging (MRI)
* Prior or concurrent therapy with SSA is permitted; a stable dose at least 2 months prior to study start and must continue on the stable dose while receiving study treatment; SSA is not considered as a systemic treatment.
* WHO PS ≤ 1
* Adequate bone marrow function or organ function

Exclusion Criteria:

* Previous treatment with any PI3K or AKT inhibitor
* Discontinuation prior mTOR inhibitor therapy due to toxicity
* Poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid, goblet cell carcinoid and small cell carcinoma
* Radiotherapy, or major surgery within 4 weeks prior to study treatment start
* Hepatic artery embolization or cryoablation/ radiofrequency ablation of hepatic metastasis within 2 months of study treatment start.
* More than 3 prior systemic treatment regimens (including cytotoxic chemotherapy, targeted therapy, immunotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (4):
  - Indiana University SC, Indianapolis, Indiana
  - Dana Farber Cancer Institute GastrointestionalCancer Clinic, Boston, Massachusetts
  - Montefiore Medical Center SC-2, The Bronx, New York
  - Ohio State Comprehensive Cancer Center/James Cancer Hospital SC, Columbus, Ohio
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Leuven, Belgium
- France (2):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Villejuif
- Novartis Investigative Site, Essen, Germany
- Italy (2):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
- Novartis Investigative Site, Rotterdam, Netherlands
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
- Novartis Investigative Site, Manchester, United Kingdom

REFERENCES:
- [Derived] Fazio N, Buzzoni R, Baudin E, Antonuzzo L, Hubner RA, Lahner H, DE Herder WW, Raderer M, Teule A, Capdevila J, Libutti SK, Kulke MH, Shah M, Dey D, Turri S, Aimone P, Massacesi C, Verslype C. A Phase II Study of BEZ235 in Patients with Everolimus-resistant, Advanced Pancreatic Neuroendocrine Tumours. Anticancer Res. 2016 Feb;36(2):713-9. PMID 26851029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase II, two-stage, multicenter study, where Stage 1 was a singlearm,open label design and Stage 2 was planned to be a randomized, double-blind study.
  However, at the end of Stage 1, the futility was met and hence the Stage 2 was not initiated.
Pre-assignment Details: Initially , the patients were started at BEZ235 400mg bid dose regimen. The preliminary safety & tolerability data fro first 3 patients treated at this dose showed all patients reported AEs leading to dose interruption. It was decided to decrease the dose of BEZ235 to 300mg bid dose regimen.
Groups:
- BEZ235 300 mg: Oral BEZ235 300 mg bid was investigated in stage 1 of study
- BEZ235 400 mg Bid: Oral BEZ235 400 mg bid was investigated in stage 1 of study
Period: Overall Study
Arm/Group | BEZ235 300 mg | BEZ235 400 mg Bid
Started | 20 | 11
Completed | 0 | 0
Not Completed | 20 | 11
Not completed — Adverse Event | 6 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Progressive disease | 12 | 4
Not completed — Study terminated by sponsor | 0 | 1
Not completed — Subject/guardian decision | 0 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of study treatment (Stage 1). This set was known as 'Analysis Set Stage 1' (AS1).
Groups:
- BEZ235 300 mg/400 mg Bid: Oral BEZ235 300 mg/400 mg bid was investigated in stage 1 of study
Arm/Group | BEZ235 300 mg/400 mg Bid
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Stage 1 - Progression Free Survival (PFS) Rate Analysis at 16 Weeks as Per Local Radiology Review
Description: PFS rate at 16 weeks was defined as a binary variable. Patients were considered as 'progression free' after 16 weeks if they had an overall lesion response of complete response (CR) partial response ('PR) or stable disease (SD)' and "progressed" if they had an overall lesion response of 'Progressive disease (PD) at the scan which occurred on day 105 after start of treatment, or later. Patients whose 16 weeks tumor assessment was unknown, missing or outside the window was not considered as 'progression free' and was considered a "failure" and counted only in the denominator for the estimation of the 16 week progression free rate.
Time Frame: 16 weeks after the first BEZ235 administration.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BEZ235 300 mg/400 mg Bid
Number analyzed (Participants) | 31
Percentage of participants | 51.6 [35.7 to 67.3]

2. Secondary Outcome: Stage 1- Overall Response Rate (ORR)
Description: Overall Response rate was defined as the proportion of patients with a best overall response of complete response or partial response, based on investigator's assessment as per RECIST criteria version 1.1. Based on futility analysis conducted at the end of stage 1, stage 2 was not initiated.
Time Frame: Baseline, every 8 weeks up to 31 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | BEZ235 300 mg/400 mg Bid
Number analyzed (Participants) | 31
Percentage of participants
  Complete response | 0.0
  Partial response | 0.0

3. Secondary Outcome: Stage 1 - Disease Control Rate
Description: Disease control rate was defined as the proportion of patients with a best overall response of Complete Response, Partial response, or Stable disease, based on the investigator's assessment per RECIST version 1.1. Based on futility analysis conducted at the end of stage 1, stage 2 was not initiated.
Time Frame: Baseline, every 8 weeks up to 31 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BEZ235 300 mg/400 mg Bid
Number analyzed (Participants) | 31
Percentage of participants | 71.0 [54.8 to 83.9]

ADVERSE EVENTS:
Groups:
- BEZ235 300 mg Bid: BEZ235 300 mg bid
- BEZ235 400 mg Bid: BEZ235 400 mg bid
Arm/Group | BEZ235 300 mg Bid | BEZ235 400 mg Bid
Serious Adverse Events (participants affected / at risk) | 8/20 | 5/11
Other Adverse Events (participants affected / at risk) | 20/20 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BEZ235 300 mg Bid (N=20) | BEZ235 400 mg Bid (N=11)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 0
LEFT VENTRICULAR HYPERTROPHY (Cardiac disorders) | 0 | 1
SYSTOLIC DYSFUNCTION (Cardiac disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 0
PYREXIA (General disorders) | 1 | 0
CHOLESTASIS (Hepatobiliary disorders) | 0 | 1
HEPATIC PAIN (Hepatobiliary disorders) | 0 | 1
ERYSIPELAS (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 2 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BEZ235 300 mg Bid (N=20) | BEZ235 400 mg Bid (N=11)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
PALPITATIONS (Cardiac disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 4
ANAL FISSURE (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 1 | 0
CHEILITIS (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 4 | 1
DIARRHOEA (Gastrointestinal disorders) | 16 | 6
DRY MOUTH (Gastrointestinal disorders) | 2 | 1
DYSPEPSIA (Gastrointestinal disorders) | 2 | 2
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
MELAENA (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 9 | 6
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 2
PROCTALGIA (Gastrointestinal disorders) | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 6 | 5
TOOTH DISCOLOURATION (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 6 | 4
ASTHENIA (General disorders) | 4 | 3
FACE OEDEMA (General disorders) | 1 | 0
FATIGUE (General disorders) | 7 | 3
INFLUENZA LIKE ILLNESS (General disorders) | 2 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 2
OEDEMA (General disorders) | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 4 | 3
PAIN (General disorders) | 0 | 1
PYREXIA (General disorders) | 4 | 1
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 | 1
HEPATIC PAIN (Hepatobiliary disorders) | 2 | 1
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 0 | 2
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 0
BRONCHITIS (Infections and infestations) | 2 | 0
CONJUNCTIVITIS (Infections and infestations) | 0 | 1
FOLLICULITIS (Infections and infestations) | 1 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 0
GINGIVITIS (Infections and infestations) | 0 | 1
INFLUENZA (Infections and infestations) | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 1 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1
ORAL HERPES (Infections and infestations) | 1 | 2
PARONYCHIA (Infections and infestations) | 1 | 0
PHARYNGITIS (Infections and infestations) | 0 | 1
RHINITIS (Infections and infestations) | 1 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 0 | 1
CONTRAST MEDIA REACTION (Injury, poisoning and procedural complications) | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 1
BLOOD CHLORIDE DECREASED (Investigations) | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 1
BLOOD IRON DECREASED (Investigations) | 1 | 0
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 | 0
BLOOD POTASSIUM INCREASED (Investigations) | 1 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 | 0
EJECTION FRACTION DECREASED (Investigations) | 1 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3 | 2
HEPATIC ENZYME INCREASED (Investigations) | 0 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 | 0
NEUTROPHIL COUNT INCREASED (Investigations) | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 2 | 2
WHITE BLOOD CELLS URINE (Investigations) | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 | 2
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 7 | 4
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCLE ATROPHY (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 0
LETHARGY (Nervous system disorders) | 0 | 2
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
MIGRAINE (Nervous system disorders) | 1 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 1
TREMOR (Nervous system disorders) | 1 | 1
AGITATION (Psychiatric disorders) | 0 | 1
DEPRESSED MOOD (Psychiatric disorders) | 0 | 1
DEPRESSION (Psychiatric disorders) | 1 | 0
HALLUCINATION (Psychiatric disorders) | 0 | 1
INSOMNIA (Psychiatric disorders) | 1 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 0
DYSURIA (Renal and urinary disorders) | 1 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 0
SCROTAL PAIN (Reproductive system and breast disorders) | 1 | 0
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 | 1
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 0 | 1
CATARRH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 1
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 | 0
HAND DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 1 | 0
NAIL TOXICITY (Skin and subcutaneous tissue disorders) | 1 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 0
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 2
RASH (Skin and subcutaneous tissue disorders) | 2 | 3
ROSACEA (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 | 1
FLUSHING (Vascular disorders) | 0 | 1
HOT FLUSH (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.